CLINICAL TRIAL: NCT00236171
Title: Evaluation of Topical Antipsoriatics in the Psoriasis Plaque Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Gottfried Wozel, MD, Technical University Dresden
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ETAPSO
Record Dates: First submitted 2005-10-04; First posted 2005-10-12 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Psoriasis Vulgaris
Keywords: topical therapy; Psoriasis Plaque Test
MeSH Terms: interventions — Tacrolimus; methylprednisolone aceponate; Blood Specimen Collection; Urinalysis; Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Protopic, Advantan
Procedure: Blood and Urine Test
Procedure: coherence tomography

SUMMARY:
The purpose of this study is to evaluate the efficacy of the topical therapies Protopic and Advantan as well as their combination against placebo in a Psoriasis Plaque Test

DETAILED DESCRIPTION:
daily psoriasis plaque tests for two weeks and optical coherence tomography (OCT) and 20-MHz-ultrasound on day 0 and day 11, 10 days post end of treatment and 20 days post end of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 Years
* Negative urine pregnancy test
* Written informed consent
* Good compliance

Exclusion Criteria:

* Patients less than 18 years
* Pregnant patients
* Patients with renal insufficiency, liver diseases
* Patients who received systemic antipsoriatic treatment or UV treatment less than 4 weeks prior to study
* Patients who used topical antipsoriatics within two weeks prior to study
* Immunosuppressed Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
sum score of psoriasis plaque tests on day 11

SECONDARY OUTCOMES:
20-MHz-ultrasound and OCT on day 11

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Wozel, Professor, Principal Investigator — Technische Universität Dresden
Locations (1):
- Technische Universität Dresden, Dresden, Saxony, Germany